CLINICAL TRIAL: NCT01514643
Title: Inflammatory Response Following Intraarticular Fracture
Acronym: PTOA
Status: Active, not recruiting | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Justin Haller, M.D., University of Utah
Other Study IDs: 51134
Record Dates: First submitted 2011-12-21; First posted 2012-01-23 (Estimated); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Intraarticular Fracture and Post-traumatic Osteoarthritis
Keywords: tibial plateau fracture; tibial plafond fracture; inflammatory cytokine profile; synovial fluid; blood serum; Post-traumatic osteoarthritis (PTOA)
MeSH Terms: conditions — Intra-Articular Fractures; Tibial Plateau Fractures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Synovial fluid and blood serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- tibial plateau or plafond fracture: Tibial plateau or plafond fracture based on radiographs and/or CT scan will have synovial fluid aspirated from both the injured and uninjured joints in either the operating room if a procedure is planned for within 24 hours or in the emergency department. While the patient is under anesthesia in the operating room, the investigators will obtain blood samples.

SUMMARY:
The purpose of the study is to investigate a relationship between the inflammatory response following intraarticular fracture and post-traumatic osteoarthritis. The investigators plan to evaluate the inflammatory cytokine profile in knee joint synovial fluid and blood serum in patients who sustain an intraarticular tibial plateau fracture and ankle joint synovial fluid and blood serum in patients who sustain an intraarticular tibial plafond fracture. This information will be combined with radiographs and patient outcome measures to determine a correlation between intraarticular inflammatory response and post-traumatic osteoarthritis.

DETAILED DESCRIPTION:
Post-traumatic osteoarthritis (PTOA) is a common cause of disability following a traumatic event involving a joint. It is estimated that PTOA may affect up to 12% of the population with symptomatic osteoarthritis, and it is associated with significant cost to the healthcare system. Given that the majority of trauma patients are younger, the impact of the condition can be particularly devastating for those in the prime of their working careers.

PTOA can develop following a variety of joint injuries, but it most predictably occurs with articular fracture. The initial traumatic injury involves a complex process of articular impaction or displacement and soft tissue disruption that leads to articular exposure to blood and marrow, a local inflammatory response, abnormal joint loading, and subsequent chondrocyte necrosis and apoptosis. However, the mechanism(s) that lead to progression from the initial injury to end-stage PTOA are largely unknown.

Inflammation can have deleterious effects on a joint. Though inflammatory cytokines have been shown to stimulate bone repair through osteoclastogenesis and recruitment of osteoblastic cells, multiple studies have demonstrated that these cytokines play a role in cartilage degradation. Increased IL-1 and TNF-a expression has been found in the cartilage of patients with osteoarthritis, and these cytokines are transiently increased after traumatic injury. Other matrix molecules including matrix metalloproteinase (MMP)-3 and cartilage oligomeric matrix protein (COMP) can be persistently elevated in synovial fluid after ACL injury.

The effect of the initial inflammatory response after intraarticular fracture on the development of PTOA remains unknown. Several authors have found elevated levels of cytokines in joints affected by trauma. However, these studies evaluated patients following an anterior cruciate ligament (ACL) injury. An intraarticular fracture likely subjects the joint to more of an inflammatory response and may place the joint at greater risk for developing osteoarthritis. There are currently no studies that link elevated levels of the inflammatory cytokines and chemokines in the setting of intraarticular trauma with PTOA. Investigating the cytokine profile in a joint immediately following intraarticular injury could lead to early targeted drug therapy with cytokine inhibitors to modify the progression of PTOA.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Radiographic evidence of tibial plateau fracture

Exclusion Criteria:

* Less than 18 years of age
* Greater than 60 years of age
* Any history of pre-existing knee osteoarthritis based on previous diagnosis or suggestive history
* Any history of autoimmune disease
* Any history of contralateral intra-articular knee injury

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients presenting with tibial plateau or plafond fracture.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2011-10; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Post-traumatic osteoarthritis (PTOA) | 2 years
  Compare mean concentrations of inflammatory cytokines profiles between each patients' injured and uninjured joints.

CONTACTS AND LOCATIONS:
Overall Officials: Justin Haller, MD, Principal Investigator — University of Utah Orthopedics
Locations (1):
- University of Utah Orthopedics, Salt Lake City, Utah, United States